CLINICAL TRIAL: NCT06503432
Title: The Effects of Programmed Death-ligand 1 on Postoperative Pain for Lung Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, director of department of Anesthesiology and Pain medicine, Peking University People's Hospital
Other Study IDs: 2020PHB252-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Postoperative Pain
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high expression of programmed death-ligand 1: According to the distribution of PD-L1 concentration levels in the plasma, participants were divided into two groups: high expression of PD-L1 (PD-L1(H)) and low expression of PD-L1 (PD-L1(L)).
- low expression of programmed death-ligand 1: According to the distribution of PD-L1 concentration levels in the plasma, participants were divided into two groups: high expression of PD-L1 (PD-L1(H)) and low expression of PD-L1 (PD-L1(L)).

SUMMARY:
The concentration of plasma programmed death-ligand 1(PD-L1) for lung cancer patients before video-assisted thoracoscopic surgery is detected. According to the distribution of plasma concentration, patients are divided into high or low expression of PD-L1. Differences in acute and chronic postoperative pain are compared between two groups of patients. And effects of PD-L1 expresion on postoperative pain in lung cancer patients are explained.

DETAILED DESCRIPTION:
Chronic pain after video-assisted thoracoscopic surgery (VATS) has been a major concern for lung cancer patients. The relationship between plasma programmed cell death ligand-1 (PD-L1) concentration and chronic pain in post-VATS is uncertain. This study aims to explore the effects of PD-L1 levels on chronic pain and provide proactive pain management regimen according to individual genetic differences.

The concentration of plasma PD-L1 for lung cancer patients before video-assisted thoracoscopic surgery is detected. According to the distribution of plasma concentration, patients are divided into high or low expression of PD-L1. Differences in acute and chronic postoperative pain are compared between two groups of patients. And effects of PD-L1 expresion on postoperative pain in lung cancer patients are explained.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status I-IV (males and females).
2. 18-80 years of age.
3. Patients undergoing video-assisted thoracoscopic surgery for malignant lung disease.

Exclusion Criteria:

1. History of opioid abuse.
2. Known psychiatric disorders.
3. Unexpected conversion to thoracotomy or transferred to intensive care unit for further treatment.
4. Combined with other surgeries or sites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent video-assisted thoracoscopic surgery for malignant lung disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the incidence of chronic pain after surgery | 3 months after surgery
  Patients were followed up by the Brief Pain Inventory questionnaire about the details of chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Tian, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China